CLINICAL TRIAL: NCT02296567
Title: Comparison of Pharmacokinetics of and Effect on Systemic Vascular Endothelial Growth Factor (VEGF) Levels Over Time of Intravitreal Ranibizumab and Bevacizumab and Aflibercept in Age Related Macular Degeneration Patients
Brief Title: Comparison of Pharmacokinetics of and Effect on Systemic VEGF Levels in Age Related Macular Degeneration Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Florida Eye Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ronald E. Frenkel, MD, Prinicipal Investigator, East Florida Eye Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ML29189
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Bevacizumab; aflibercept; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group 1 Lucentis 4 weeks (Active Comparator): Blood samples will be collected from patients receiving ranibizumab following the first dose of standard care therapy.
  Interventions: Drug: Ranibizumab
- Group 2 Avastin 4 weeks (Active Comparator): Blood samples will be collected from patients receiving bevacizumab following the first dose of standard care therapy.
  Interventions: Drug: Bevacizumab
- Group 3 Eylea 4 weeks (Active Comparator): Blood samples will be collected from patients receiving aflibercept following the first dose of standard care therapy.
  Interventions: Drug: Aflibercept
- Group 4 Lucentis 6 weeks (Active Comparator): Blood samples will be collected from patients receiving ranibizumab following the first dose of standard care therapy.
  Interventions: Drug: Ranibizumab
- Group 5 Avastin 6 weeks (Active Comparator): Blood samples will be collected from patients receiving bevacizumab following the first dose of standard care therapy.
  Interventions: Drug: Bevacizumab
- Group 6 Eylea 6 weeks (Active Comparator): Blood samples will be collected from patients receiving aflibercept following the first dose of standard care therapy.
  Interventions: Drug: Aflibercept
- Group 7 Lucentis 8 weeks (Active Comparator): Blood samples will be collected from patients receiving ranibizumab following the first dose of standard care therapy.
  Interventions: Drug: Ranibizumab
- Group 8 Avastin 8 weeks (Active Comparator): Blood samples will be collected from patients receiving bevacizumab following the first dose of standard care therapy.
  Interventions: Drug: Bevacizumab
- Group 9 Eylea 8 weeks (Active Comparator): Blood samples will be collected from patients receiving aflibercept following the first dose of standard care therapy.
  Interventions: Drug: Aflibercept
- Group 10 Control Group no treatment (Active Comparator): Blood samples will be collected from patients who are not receiving anti-VEGF treatment.
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Ranibizumab — Drug: Ranibizumab Subjects will receive intravitreal Ranibizumab as part of their routine medical care.
  Other Names: Lucentis
  Arms: Group 1 Lucentis 4 weeks
Drug: Bevacizumab — Drug: Bevacizumab Subjects will receive intravitreal Bevacizumab as part of their routine medical care.
  Other Names: Avastin
  Arms: Group 2 Avastin 4 weeks
Drug: Aflibercept — Drug: Aflibercept Subjects will receive intravitreal Aflibercept as part of their routine medical care.
  Other Names: Eylea
  Arms: Group 3 Eylea 4 weeks
Drug: Ranibizumab — Drug: Ranibizumab Subjects will receive intravitreal Ranibizumab as part of their routine medical care.
  Other Names: Lucentis
  Arms: Group 4 Lucentis 6 weeks
Drug: Bevacizumab — Drug: Bevacizumab Subjects will receive intravitreal Bevacizumab as part of their routine medical care
  Other Names: Avastin
  Arms: Group 5 Avastin 6 weeks
Drug: Aflibercept — Drug: Aflibercept Subjects will receive intravitreal Aflibercept as part of their routine medical care
  Other Names: Eylea
  Arms: Group 6 Eylea 6 weeks
Drug: Ranibizumab — Drug: Ranibizumab Subjects will receive intravitreal Ranibizumab as part of their routine medical care
  Other Names: Lucentis
  Arms: Group 7 Lucentis 8 weeks
Drug: Bevacizumab — Drug: Bevacizumab Subjects will receive intravitreal bevacizumab as part of their routine medical care
  Other Names: Avastin
  Arms: Group 8 Avastin 8 weeks
Drug: Aflibercept — Drug: Aflibercept Subjects will receive intravitreal Aflibercept as part of their routine medical care
  Other Names: Eylea
  Arms: Group 9 Eylea 8 weeks
Other: Control Group — Control group Subjects will no previous anti-VEGF treatment
  Arms: Group 10 Control Group no treatment

SUMMARY:
To demonstrate the effects of Lucentis (ranibizumab), Avastin ( bevacizumab), and Eylea ( aflibercept) on the levels of naturally occurring Vascular Endothelial Growth Factor (VEGF) in the systemic circulation of Age Related Macular Degeneration patients currently treated with these medications.

DETAILED DESCRIPTION:
To determine plasma levels of VEGF and serum Pharmacokinetic (PK) levels after varying lengths of time following intravitreal injection with Avastin, Lucentis, or Eylea in exudative macular degeneration. Patients will be tested while following a normal course of treatment in our institute. All screenings and testing will be conducted in three study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent for participation in this study.
2. Adults ≥ 50 years of age with exudative macular degeneration treated with Avastin, Lucentis, or Eylea in previously determined time intervals exclusive to a single anti-VEGF treatment type for not than three months.
3. CONTROL GROUP: Age matched control group with no previously diagnosed exudative macular degeneration will also be enrolled.
4. Provide signed informed consent.

Exclusion Criteria:

1. Uncontrolled blood pressure (defined as systolic > 160mm Hg or Diastolic > 95mm Hg while patient is sitting)
2. Uncontrolled diabetes mellitus defined by Hemoglobin A1c (HbA1C > 12% at screening)
3. Concomitant ocular or systemic administration of drugs that may interfere with or potentiate the mechanism of action of anti-VEGF medications.
4. Previous administration of systemic anti-angiogenic medications within 3 months
5. Participation in a simultaneous medical investigation or trial.
6. Treatment within 2 months with anti-VEGF agent in the fellow eye or anticipated need for further treatment during the study.
7. Patients with any cancer diagnosis in remission for less than five years with the exception that patients with skin cancers, basal cell or squamous cell, treated exclusively or topical treatment will be allowed.
8. Female patients who have not reached menopause, defined as cessation of menses for a minimum of twelve months with no perimenopausal symptoms.
9. Patients who have significant wound healing during the trial.
10. Patients with a history of vitrectomy in the study eye.
11. patients with uncontrolled psoriasis, rheumatoid arthritis, osteoarthritis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in serum and plasma levels of free Vascular Endothelial Growth Factor | up to 8 weeks
  Serum and plasma levels of free vascular endothelial growth factor will be measured up to 8 weeks following the standard of care treatment.

SECONDARY OUTCOMES:
Change in Serum drug levels in nanomoles (nM) units following treatment | 8 weeks
  Serum levels of Ranibizumab, Bevacizumab, or Aflibercept will be measured up to 8 weeks following the standard of care treatment.
Amount of fluid (cubic mm) as measured by Ocular Coherence Tomography in the contralateral eye will be correlated with systemic Vascular Endothelial Growth Factor levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Frenkel, MD, Principal Investigator — East Florida Eye Institute
Locations (1):
- East Florida Eye Institute, Stuart, Florida, United States